CLINICAL TRIAL: NCT04350086
Title: Prospective Study of the Use of Dexmedetomidine in Light to Moderate Sedation in the Patient in the Palliative Situation of a Sars-cov-2 / COVID-19 Infection
Brief Title: Use of Dexmedetomidine in Light to Moderate Sedation in the Patient in the Palliative Situation of a Sars-cov-2 / COVID-19 Infection
Acronym: PRODEX
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: unfavorable opinion of the ethics committee
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 87RI20_0011 (PRODEX)
Record Dates: First submitted 2020-04-13; First posted 2020-04-16 (Actual); Last update posted 2020-09-02 (Actual); Status verified 2020-04

CONDITIONS: COVID-19 Infection; Sars-cov-2; Respiratory Failure; Palliative Situation
Keywords: COVID-19; sars-cov-2; infection; respiratory failure; palliative situation
MeSH Terms: conditions — COVID-19; Respiratory Insufficiency; Infections | interventions — Therapeutics; Dexmedetomidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental arm (Experimental)
  Interventions: Drug: Treatment with Dexmedetomidine

INTERVENTIONS:
Drug: Treatment with Dexmedetomidine — Administration of Dexmedetomidine in continuous infusion by electric syringe pump at a dose of 0.4 µg / kg / h, with dose adjustment according to the sedation score and tolerance.

SUMMARY:
The current sars-cov-2 epidemic is responsible for severe respiratory infections leading to end-of-life situations.

Dexmedetomidine may be indicated in mild to moderate sedation in palliative patients, due to its pharmacological characteristics.

The hypothesis of this study is that Dexmedetomidine would allow effective and safe light sedation in patients with respiratory failure in palliative situations suffering from Covid-19 infection.

ELIGIBILITY:
Inclusion Criteria:

1. Major patient
2. Relating to palliative care
3. With sars-cov-2 infection
4. Requiring light to moderate sedation corresponding to a RASS score of -1 to -3

Exclusion Criteria:

1. Pregnant, lactating woman.
2. Hypersensitivity to the active substance or to any of the excipients listed in section 6.1 of the summary of product characteristics
3. Advanced heart block (level 2 or 3) unless a pacemaker.
4. Uncontrolled hypotension.
5. Acute cerebrovascular pathologies.
6. Use of other sedative drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-04-20 (Estimated); Primary Completion 2020-11-20 (Estimated); Study Completion 2020-11-20 (Estimated)

PRIMARY OUTCOMES:
Efficacy of mild to moderate palliative sedation induced by Dexmedetomidine. | Day 30
  Number of days of mild to moderate sedation induced by dexmedetomidine until death or change of molecule.

SECONDARY OUTCOMES:
Overall survival of patients on Dexmedetomidine | Day 30
  Overall survival time in days from inclusion.
Daily analgesic effect of Dexmedetomidine | Day 30
  The daily effectiveness of Dexmedetomidine on pain assessed by the NCS-R scale (Nociception Coma Scale) : the score is between 0 and 9.
Other sedative pharmacological agents | Day 30
  Number of the various sedative molecules used in the subjects of the study in addition to Dexmedetomidine.
Average dosage required for Dexmedetomidine to achieve mild to moderate sedation | Day 30
  Daily dosage measurement in ug / kg / h of Dexmedetomidine necessary to obtain light to moderate sedation

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital, Limoges, France

IPD SHARING:
Plan to Share IPD: No